CLINICAL TRIAL: NCT00886847
Title: Specimen Adequacy and Diagnostic Agreement of Fine Needle Aspiration (FNA) VS. Fine Needle Capillary Sampling (FNC) of Endobronchial Ultrasound-Guided Biopsy of Mediastinal Lymph Nodes
Brief Title: Comparison of Endobronchial Ultrasound-Guided Biopsy Using Fine Needle Aspiration Versus Fine Needle Capillary Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-0051
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-08

CONDITIONS: Lymphadenopathy
Keywords: Lung; Lymphadenopathy; Enlarged hilar or/and mediastinal lymph adenopathy; Benign; Malignant; Mediastinal lymph nodes; Hilar lymph nodes; Fine Needle Aspiration; FNA; Fine Needle Capillary Sampling; FNC; Endobronchial Ultrasound-Guided Biopsy; EBUS; Tissue Sample; Suction
MeSH Terms: conditions — Lymphadenopathy | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBUS FNA vs FNC (Experimental)
  Interventions: Procedure: Lymph Node Needle Tissue Collections

INTERVENTIONS:
Procedure: Lymph Node Needle Tissue Collections — Total of two lymph nodes sampled per patient. Four biopsies will be taken from each lymph node. Two with suction (FNA) and two without suction (FNC).
  Other Names: Fine Needle Aspiration; Fine Needle Capillary

SUMMARY:
Primary objective:

* To estimate the degree of agreement in diagnosis of cytologic samples from mediastinal lymph nodes obtained by Endobronchial Ultrasound (EBUS)-guided Fine Needle Capillary Sampling (FNC) versus Fine Needle Aspiration (FNA).

Secondary objective:

* To compare the quality of cytologic samples from mediastinal lymph nodes obtained by EBUS-guided FNC versus FNA. The quality of the samples will be assessed initially by MDACC on-site cytology technicians, and then corroborated by physicians in the department of cytology. This assessment will be performed utilizing the Mair's score 3. The score consists of a 0-10 scale: 1-2= poor; 3-6=good; 7-10=superior.

DETAILED DESCRIPTION:
Tissue Sample Collection:

If you agree to take part in this study, you will have your already scheduled endobronchial ultrasound-guided biopsy performed after you have been given a drug to make you sleep. You will be asked to sign a separate informed consent for the biopsy procedure.

During a standard of care biopsy procedure, there are normally 3-5 tissue sample collections performed. For the purposes of this study, you will have a total of 4 tissue collections performed during the biopsy procedure. Two tissue collections (2) using the FNC method, and 2 tissue collections using the FNA method.

If the first 4 tissue sample collections do not provide good enough tissue samples to perform the diagnosis, additional sample collections may be performed. If more samples are collected, these samples will not be used for the purposes of this study and will only be collected for diagnostic purposes.The sampling will be done by the pulmonologist who is performing your procedure.

The first 4 tissue samples that are collected for the purposes of this study will be examined to determine the quality of the sample as well as for diagnostic purposes.

Medical Record Information:

Information from your medical record will be collected 1 time for this study. The information collected will include information about your diagnosis, the number of radiation treatments you may have had, and additional information about your medical history. The information will be de-identified and stored in a research database on a password protected computer that only the study doctor and study staff will have access to.

Length of Study:

You will remain on study for the duration of biopsy procedure. After the biopsy has been performed, and your medical record information has been collected you will no longer be on study.

This is an investigational study. The endobronchial ultrasound-guided biopsy of the lymph nodes is FDA approved. Both methods of tissue collection (FNA and FNC) are FDA approved for the purposes of this study.

Up to 200 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. patients 18 years or older
2. Patients in which EBUS is indicated based on the suspicion of either benign or malignant disease in mediastinal and/or hilar lymph nodes. This will include patients who are in the hospital.

Exclusion Criteria:

1. patients under 18 years or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of times FNA and FNC agree on patient diagnosis (concordance) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo C. Morice, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Casal RF, Staerkel GA, Ost D, Almeida FA, Uzbeck MH, Eapen GA, Jimenez CA, Nogueras-Gonzalez GM, Sarkiss M, Morice RC. Randomized clinical trial of endobronchial ultrasound needle biopsy with and without aspiration. Chest. 2012 Sep;142(3):568-573. doi: 10.1378/chest.11-0692. PMID 22156610
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org